CLINICAL TRIAL: NCT06726642
Title: CfDNA in Hereditary And High-risk Malignancies (CHARM) 2: Evaluating the Performance of a cfDNA Blood Test for Early Cancer Detection
Brief Title: CfDNA in Hereditary And High-risk Malignancies 2
Acronym: CHARM2
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: British Columbia Cancer Agency (Other); Eastern Health (Other); IWK Health Centre (Other); Jewish General Hospital (Other); Sinai Health System (Other); The Hospital for Sick Children (Other); University of Alberta (Other); Women's College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5766
Record Dates: First submitted 2024-11-08; First posted 2024-12-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Cancer Syndrome
Keywords: cfDNA; cell-free DNA; Hereditary cancer syndrome; BRCA1; BRCA2; Lynch Syndrome; Hereditary breast and ovarian cancer (HBOC); Liquid biopsy; Circulating tumor DNA; Hereditary Diffuse Gastric Cancer (HDGC); Li-Fraumeni syndrome
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary Breast and Ovarian Cancer Syndrome; Stomach Neoplasms; Li-Fraumeni Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma and buffy coat samples, and/or DNA extracted from blood plasma and buffy coat samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test cohort: All participants in the experimental cohort will provide blood samples tri-annually (every 4 months) for 4 years, either at the study hospital or at a local blood laboratory (e.g., LifeLabs). Whenever possible, patients will have research blood collected at the same time as routine blood collections for clinical purposes to avoid additional venipunctures. The samples will undergo cfDNA analysis and all results will be returned to participants by the study team. Participants who receive a "positive" cfDNA assay result will be offered follow-up diagnostic procedures to confirm or rule out the presence of a malignancy. Participants will also complete questionnaires and semi-structured interviews to explore their experience with cfDNA testing and understand perceptions of the clinical utility of cfDNA tests for HCS management.
  Interventions: Diagnostic Test: Cell-free DNA analysis
- Control: Participants in the control cohort will not receive the cfDNA blood test and will continue to receive standard-of-care cancer surveillance according to current guidelines, as they were prior to study enrollment. Participants will complete questionnaires and semi-structured interviews to explore their experience with cfDNA testing and to understand their perception of the clinical utility of cfDNA tests for HCS management.

INTERVENTIONS:
Diagnostic Test: Cell-free DNA analysis — Analysis of cell-free DNA in blood plasma will involve targeted sequencing of key cancer-related genes, cell-free methylated DNA immunoprecipitation and high-throughput sequencing (cfMeDIP-seq), and shallow whole genome sequencing (sWGS).
  Groups: Test cohort

SUMMARY:
The goal of this study is to understand the performance of an experimental blood test that aims to detect early tumors in patients with hereditary cancer syndromes. If this new blood test is accurate, it could be used to screen patients for cancer and allow for earlier cancer detection. The study will compare cancer detection rates between those receiving the new blood test and those receiving standard care, assess if the test leads to earlier cancer diagnosis, and evaluate its impact on patient outcomes. The study will also use questionnaires and interviews to understand how patients feel about the blood test, its incorporation into routine medical care, and perceptions of the medical value of test results. This research could lead to more effective and less invasive cancer screening for high-risk individuals.

DETAILED DESCRIPTION:
Through the CHARM Consortium (www.charmconsortium.ca), the investigators have shown that cell-free DNA (cfDNA) profiling can enable more frequent cancer surveillance from readily accessible blood collections. The investigators are now conducting a prospective, multi-center, randomized control trial of cfDNA testing of 1,000 HCS carriers from across Canada to 1) compare cancer detection rates with and without cfDNA testing, 2) assess cancer stage shift and clinical impact reducing mortality and morbidity cancers, and 3) assess impact of access to cfDNA results on patients' quality of life and psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of hereditary breast and ovarian cancer (HBOC), Lynch Syndrome (LS), Neurofibromatosis type I (NF1), Li-Fraumeni Syndrome (LFS), PALB2, and Hereditary Diffuse Gastric Cancer (HDGC), (i.e., patients with an identified pathogenic variant in the respective cancer predisposition gene, or patients with uninformative genetic testing but with a family history suggestive of the cancer predisposition syndrome).
* Patients must be receiving standard-of-care clinical assessment for cancer by a managing physician under a provincial screening program or cancer surveillance protocol.
* All patients must have signed and dated an informed consent form for this study.

Exclusion Criteria:

* Patients must not have a personal history of cancer diagnosed and treated within 3 years prior to the expected first sample collection date for this study. If a patient has a personal history of cancer, treatment must have been completed successfully at least 3 years prior to first study sample collection.
* Patients diagnosed more than 3 years prior to the expected first sample collection date, but never been treated for the cancer.
* Patients undergoing investigations for a clinical suspicion of cancer.
* Patients who are not able to comply with the protocol (i.e., tri-annual blood sample collection if randomized into the experimental cohort).

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population to be studied includes:
  Any individual that underwent clinical genetic testing for hereditary breast and ovarian cancer syndrome, Lynch Syndrome, Neurofibromatosis Type 1, Li-Fraumeni Syndrome or Hereditary Diffuse Gastric Cancer, and was found to carry a detectable variant that is likely pathogenic or pathogenic.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Determine the cancer detection rate of the cfDNA sequencing assay in patients with HCS. | 4 years from enrollment in the study.
  The investigators will assess the performance of the cfDNA assay for cancer detection in patients with HCS, including assay sensitivity, specificity, positive predictive value (PPV,) and negative predictive value (NPV). The test performance endpoint is a diagnosis of cancer and will be assessed at multiple points during the study (at a minimum yearly).

SECONDARY OUTCOMES:
To assess the time to cancer diagnosis using cfDNA sequencing compared to controls. | 4 years from enrollment in the study.
  The investigators will establish whether blood plasma cfDNA testing can detect cancers at the same time as, or earlier, than conventional standard-of-care screening tests for carriers of HCS. The investigators will also assess the time to disease management in carriers receiving cfDNA sequencing results compared to controls.
To assess the detection rate of cancers with no standard-of-care screening available using cfDNA sequencing. | 4 years from enrollment in the study.
  To establish whether cfDNA testing increases the frequency of cancers detected, in particular cancer types with limited detection rates using standard-of-care (e.g., pancreatic cancer, endometrial cancer).
Assess the impact of tri-annual cfDNA testing on participant cancer worry. | 4 years from enrollment in the study.
  The investigators will assess the impact of tri-annual cfDNA testing on participants' cancer related worry, using the Cancer Worry Scale (PMID: 19382100).
Assess the impact of tri-annual cfDNA testing on cancer risk perception. | 4 years from enrollment in the study.
  The investigators will assess the impact of tri-annual cfDNA testing on participants' risk perception, using the Multidimensional Impact of Cancer Risk Assessment (PMID: 12433008).
Assess the impact of tri-annual cfDNA testing on cancer anxiety and depression. | 4 years from enrollment in the study.
  The investigators will assess the impact of tri-annual cfDNA testing on participants' anxiety and depression using the Hospital Anxiety and Depression Scale (PMID: 18325093).

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kim, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (8):
- Canada (8):
  - BC Cancer Agency, Vancouver, British Columbia
  - Eastern Health, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farncombe KM, Wong D, Norman ML, Oldfield LE, Sobotka JA, Basik M, Bombard Y, Carile V, Dawson L, Foulkes WD, Malkin D, Karsan A, Parkin P, Penney LS, Pollett A, Schrader KA, Pugh TJ, Kim RH; CHARM consortium. Current and new frontiers in hereditary cancer surveillance: Opportunities for liquid biopsy. Am J Hum Genet. 2023 Oct 5;110(10):1616-1627. doi: 10.1016/j.ajhg.2023.08.014. PMID 37802042
- See also: CHARM consortium website — https://charmconsortium.ca/about/